CLINICAL TRIAL: NCT06847620
Title: Evaluation of the Effect of Verapamil When Added to Bupivacaine in Ultrasound-guided Supraclavicular Block in Hand Surgeries
Brief Title: Effect of Verapamil as an Adjuvant to Local Anaethetics in Supraclav Block for Hand Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FMASU MS165/2024
Record Dates: First submitted 2025-01-05; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-02

CONDITIONS: Hand Surgery
MeSH Terms: interventions — Bupivacaine; Single Person; Verapamil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- • Group A (the control group) (Active Comparator): group A: will receive 20 ml of plain bupivacaine 0.25% (equivalent to 50 mg) plus 2 ml of normal saline.
  Interventions: Procedure: Supraclavicular Brachial Plexus Block; Drug: Bupivacaine 0.25% 20ml alone
- Group B (Active Comparator): Group B : will receive 20 ml of bupivacaine 0.25% (equivalent to 50 mg) plus 2 ml verapamil (equivalent to 5 mg)
  Interventions: Procedure: Supraclavicular Brachial Plexus Block; Drug: bupivacaine 0.25% And verapamil

INTERVENTIONS:
Procedure: Supraclavicular Brachial Plexus Block — The block will be performed using a portable ultrasound system (sonosite M-turbo USA) with linear high-frequency transducer (12HZ) to get the sonographic anatomy of brachial plexus in the transverse and longitudinal planes.
Drug: Bupivacaine 0.25% 20ml alone — will receive 20 ml of plain bupivacaine 0.25% (equivalent to 50 mg) plus 2 ml of normal saline.
  Arms: • Group A (the control group)
Drug: bupivacaine 0.25% And verapamil — will receive 20 ml of bupivacaine 0.25% (equivalent to 50 mg) plus 2 ml verapamil (equivalent to 5 mg
  Arms: Group B

SUMMARY:
The aim of this study is to evaluate the role of verapamil when added to bupivacaine in ultrasound-giuded supraclavicular Brachial plexus block regarding the duration of action of the block, onset of action and the need of rescue analgesia.

DETAILED DESCRIPTION:
Preoperative Period All patients will clinically be assessed and routine preoperative investigations will be done: Complete blood picture, Coagulation profile, liver function tests, kidney function tests, fasting blood sugar and ECG. The initial vital data will be measured after applying the standard monitoring including pulse oximetry, non-invasive blood pressure and ECG. All patients will be admitted after fasting for 6 hours.

Intraoperative Period On arrival of the patients to the operative room, electrocardiography, non-invasive blood pressure, and pulse oximetry will be applied. Baseline parameters such as systolic blood pressure (SBP), diastolic blood pressure (DBP), mean blood pressure (MBP), heart rate (HR), and oxygen saturation (SpO2) will be recorded. Intravenous (IV) line will be inserted and IV lactated Ringer will be started.

The block will be performed using a portable ultrasound system (sonosite M-turbo USA) with linear high-frequency transducer (12HZ) to get the sonographic anatomy of brachial plexus in the transverse and longitudinal planes.

Under aseptic conditions, the ultrasound probe will be situated parallel to the clavicle in the supraclavicular area to show the plexus as a "bunch of grapes" or as having a "honeycomb" appearance. The block will be done with a short beveled echogenic needle 5 cm, 22 G for optimal control and visibility. The predetermined volume of 22 ml will be injected around the brachial plexus after negative aspiration to avoid inadvertent intravascular injection keeping in mind adequate block of lower trunk. Distension of brachial plexus sheath will be regarded as an indication of successful block "Donut sign". A massage for 5 min will be applied to aid an equal volume distribution.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 21-70 years old
* Patients with ASA I / II
* patients undergoing hand surgeries

Exclusion Criteria:

* Patients refusal
* Skin infection at the injection site.
* Contraindications to regional anaesthesia as bleeding disorders
* Allergy to bupivacaine or other drugs involved in the study.
* Uncooperative patients.
* BMI >35
* Patients taking medications for psychiatric illness

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2024-10-15 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure | The duration from giving the block till the need of rescue analgesia in post op 24 hours
  Duration between performing the block and the need of rescue analgesia in patients receiving ultrasound-guided supraclavicular Brachial plexus block with bupivacaine as sole agent versus bupivacaine and verapamil.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Before 2/2025
Access Criteria: Free